CLINICAL TRIAL: NCT02602054
Title: The Best Treatment Strategy: Surgical Versus Pharmacological, to Close the Ductus Arteriosus Persistent in Preterm Infants. A Randomized Controlled Trial
Brief Title: The Best Treatment Strategy: Surgical vs Pharmacological to Close the Ductus Arteriosus Persistent in Preterm Infants
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General Naval de Alta Especialidad - Escuela Medico Naval (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HGNAE-07
Record Dates: First submitted 2015-11-08; First posted 2015-11-11 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Persistent Ductus Arteriosus
Keywords: persistent ductus arteriosus; preterm infants; surgical treatment; pharmacological treatment
MeSH Terms: conditions — Ductus Arteriosus, Patent | interventions — Surgical Procedures, Operative; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgical treatment (Experimental): Implement surgical treatment for closure of patent ductus arteriosus
  Interventions: Procedure: Surgical treatment
- Control group (Active Comparator): - Indomethacin: Administer 1 full cycle (3 doses) of indomethacin (1 dose every 12 hours) for 2 days Dose 0.1 - 0.25 mg / kg
  - Ibuprofen: Administer 1 full cycle (3 doses) of ibuprofen (1 dose every 24 hours) for 2 days Dose 05 - 10 mg / kg
  - Acetaminophen: Administer 1 full cycle (12 doses) of acetaminophen (1 dose every 6 hours) for 3 days Dose 15 mg / kg
  Interventions: Drug: Control group

INTERVENTIONS:
Procedure: Surgical treatment — Standard left thoracotomy
  Other Names: Surgery
  Arms: Surgical treatment
Drug: Control group — - Indomethacin:
  Administer 1 full cycle (3 doses) / (1 dose every 12 hours) in the first fourteen days of life:
  Preterm infants less than 48 hours of life: first dose 0.2 mg/kg, second dose 0.1 mg/kg and third dose 0.1 mg/kg Preterm infants more than 48 hours of life: first dose 0.2 mg/kg, second dose 0.2 mg/kg and third dose 0.2 mg/kg And preterm infants more than 7 days of life: first dose 0.2 mg/kg, second dose 0.25 mg/kg and third dose 0.25 mg/kg - Ibuprofen:
  Administer 1 full cycle (3 doses) / (1 dose every 24 hours) in the first fourteen days of life of preterm infants:
  First dose 10 mg/kg Second dose 05 mg/kg Third dose 05 mg/kg
  - Acetaminophen
  Administer 1 full cycle, in the first fourteen days of life in preterm infants:
  Acetaminophen 15 mg/kg every 6 hours for 3 days
  Other Names: Pharmacological
  Arms: Control group

SUMMARY:
The decision to treat patent ductus arteriosus in preterm infants, varies from a conservative, medical or immediate surgical treatment; although, at present, there is some controversy about this decision. This study aims to determine the efficacy and safety of surgical versus pharmacological treatment of patent ductus arteriosus in preterm infants.

DETAILED DESCRIPTION:
The ductus arteriosus varies in length, diameter and morphology. The duct closure occurs in two stages: the first one or functional closure; the second or anatomical closure. This condition is associated with other heart diseases, which modify the natural history and require individualized treatment. Treatment varies from conservative, pharmacological or surgical treatment, and there are many controversies regarding the treatment decision. And aims of the closure, is to decrease the likelihood of irreversible pulmonary vascular disease, reduce associated morbidity and mortality. The role of prostaglandin E2 is the permeability of the conduit, by which is indicated the use of cyclooxygenase inhibitors for closure (indomethacin and ibuprofen). In various research studies many factors associated with failure of pharmacological treatment (gestational age, antenatal indomethacin less than 48 hours before delivery, use of high frequency ventilation) are reported, therefore, there is an alternative treatment which is surgical closure. In the pharmacological treatment of ductus arteriosus persistent it should be individualized according to gestational age, respiratory condition and size of the newborn. With early drug treatment can achieve closure of patent ductus arteriosus in up to 90% of cases, while the late treatment between 50-65%. However, it is reported that after treatment with indomethacin, reopening occurs, two doses are recommended more after the first, in addition to its side effects, contraindications and complications. As well, ibuprofen contraindications. So the closure of the ductus arteriosus persistent may be performed by hemodynamics and surgical closure (standard left thoracotomy or thoracoscopic technique). There are specific indications for surgical treatment (no response to two cycles of medical treatment in newborns with less than 1000 gr weight in which I fail one indomethacin, absolute contraindications to it, with significant hemodynamic repercussions. With surgical treatment before the third week of life minimizing morbidity. it is reported by many authors that complications are rare and mortality is associated with other complications of prematurity. So Surgical treatment is considered as an alternative because of its low incidence of complications, mortality and lower cost, plus a total occlusion between 94-100% Because of this, the treatment of patent ductus arteriosus in preterm infants, ranging from conservative treatment, medical or surgical, and currently there is much controversy in the treatment decision.

This study aims to determine the efficacy and safety of surgical versus pharmacological treatment for the permanent closure of the patent ductus arteriosus in preterm infants.

Methods: Is open label randomized controlled the clinical trial with: 1) experimental group assigned to surgical treatment; 2) control group assigned to pharmacological treatment, for closure of patent ductus arteriosus.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants
* Preterm infants hospitalized in the Neonatal Intensive Care Unit with a diagnosis of patent ductus arteriosus

Exclusion Criteria:

* Preterm infants with supportive treatment and / or drug prior to patent ductus arteriosus in another medical unit
* Preterm infants diagnosed with heart disease associated complex.
* Preterm infants with associated disease (not hemodynamic or cardiovascular) and its impact on his state of health prior to drug treatment and / or surgery
* Preterm infants with contraindications to pharmacological and / or surgery treatment
* Newborns diagnosed with patent ductus arteriosus but with incomplete medical records

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-04 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Success rate of closure patent ductus arteriosus | 10 days after treatment
  Tracking each patient for 10 days after treatment (surgical / pharmacological) to verify success rate of closure of patent ductus arteriosus (Failure of ductal closure ) (%)

SECONDARY OUTCOMES:
Time from diagnosis to resolution of patent ductus arteriosus | 1 month
  To compare the time from diagnosis to resolution of patent ductus arteriosus (days)
Time from start of treatment until resolution | 10 days after treatment
  To compare the time from start of treatment until resolution of patent ductus arteriosus (days)
Time limitation of family contact | 1 month
  To compare the time limitation of family contact from diagnosis to hospital discharge of newborns of patent ductus arteriosus (days)
Adverse effects and complications of treatment | 10 days
  Describe the type of adverse effects and / or complications (Chronic lung disease , Intraventricular haemorrhage, Creatinine level > 1.8 mg/dl, Pneumothorax , Sepsis, Necrotising enterocolitis, Retinopathy of prematurity, Other bleeding) and the frequency of the two study groups (yes / no)
Death before discharge | 1 month
  To compare related mortality among surgical and pharmacological treatment (%)
Time of mechanical ventilatory support, parenteral nutrition, fasting, supplementary O2 | 1 month
  To compare the duration of mechanical ventilatory support, parenteral nutrition, fasting, supplementary O2 (days).
Anatomy of the ductus arteriosus persistent | 1 month
  Describe the size of the ductus arteriosus (mm)
Gestational age at birth | At birth
  Describe the gestational age of neonates (weeks)
Apgar | At birth
  Describe the Apgar score of newborns (3-9)
Blood flow | 1 month
  Describe the direction of blood flow of the ductus arteriosus (left-right, left-right, two-way)
Gradient of the ductus arteriosus | 1 month
  Describe the gradient of the ductus arteriosus (mmHg).

CONTACTS AND LOCATIONS:
Overall Officials: Esaú Luis Nieto, Pediatrician, Principal Investigator — Hospital General Naval de Alta Especialidad - Escuela Medico Naval
Locations (1):
- Hospital General Naval de Alta Especialidad, Distrito Federal, Mexico City, Mexico

REFERENCES:
- [Result] Gallardo MAF, González SJM, et al. Experiencia en el cierre quirúrgico de ducto arterioso permeable en la Unidad de Cuidados Intensivos Neonatales de un hospital de segundo nivel en Guadalajara, Jalisco, México. Bol Med Hosp Infant Mex 2010; 67: 128-32
- [Result] Staines OH, Fuentes TMA, Staines AR. Tratamiento quirúrgico del conducto arterioso persistente. Rev Mex Cir Ped 2005; 12: 39-45.
- [Result] Golombek SG, Sola A, Baquero H, Borbonet D, Cabanas F, Fajardo C, Goldsmit G, Lemus L, Miura E, Pellicer A, Perez JM, Rogido M, Zambosco G, van Overmeire B; Primer Grupo de Consenso Clinico SIBEN. [First SIBEN clinical consensus: diagnostic and therapeutic approach to patent ductus arteriosus in premature newborns]. An Pediatr (Barc). 2008 Nov;69(5):454-81. doi: 10.1157/13128003. Spanish. PMID 19128748
- [Result] Elorza MD, Pérez RJ, Quero JJ. Tratamiento del Ductus Arterioso Persistente sintomático del recién nacido pretérmino. Hospital Universitario La Paz. Servicio Madrileño de Salud. 2005 (3): 1-8.
- [Result] Hernando BG, et al. Atención médica a niños < 30 semanas de gestación con conducto arterioso persistente. Rev Mex Pediatr. 2013; 80 (4): 131-135.
- [Result] San Luis-Miranda R, Arias-Monroy LG, Peralta-Pedrero ML, Lazaro-Castillo JL, Leon-Avila JL, Benitez-Arechiga ZM, Jauregui-Ruiz O, Yanez-Gutierrez L, Manrique-Valle M. [Clinical guide practice. Patent ductus arteriosus]. Rev Med Inst Mex Seguro Soc. 2012 Jul-Aug;50(4):453-63. Spanish. PMID 23234752
- [Result] Lee JH, Ro SK, Lee HJ, Park HK, Chung WS, Kim YH, Kang JH, Kim H. Surgical Ligation on Significant Patent Ductus Arteriosus in Very Low Birth Weight Infants: Comparison between Early and Late Ligations. Korean J Thorac Cardiovasc Surg. 2014 Oct;47(5):444-50. doi: 10.5090/kjtcs.2014.47.5.444. Epub 2014 Oct 5. PMID 25346899
- [Result] Moore GP, Lawrence SL, Maharajh G, Sumner A, Gaboury I, Barrowman N, Lemyre B. Therapeutic strategies, including a high surgical ligation rate, for patent ductus arteriosus closure in extremely premature infants in a North American centre. Paediatr Child Health. 2012 Apr;17(4):e26-31. doi: 10.1093/pch/17.4.e26. PMID 23543702
- [Result] Sung SI, Choi SY, Park JH, Lee MS, Yoo HS, Ahn SY, Chang YS, Park WS. The timing of surgical ligation for patent ductus arteriosus is associated with neonatal morbidity in extremely preterm infants born at 23-25 weeks of gestation. J Korean Med Sci. 2014 Apr;29(4):581-6. doi: 10.3346/jkms.2014.29.4.581. Epub 2014 Apr 1. PMID 24753708
- [Result] Lam JY, Lopushinsky SR, Ma IWY, Dicke F, Brindle ME. Treatment Options for Pediatric Patent Ductus Arteriosus: Systematic Review and Meta-analysis. Chest. 2015 Sep;148(3):784-793. doi: 10.1378/chest.14-2997. PMID 25835756
- [Result] Kim HK, et al. Effect of indomethacin treatment in full-term infants with symptomatic patent ductus arteriosus. Korean J Perinatol 2013; 24 (4): 237-43.
- [Result] Kwon NH, Lee JH, et al. Risk Factors of Failure of Ibuprofen Treatment in Preterm Infants with HS PDA. Korean J Perinatol 2014; 25 (4): 257-65.
- [Result] Sadeck LS, Leone CR, Procianoy RS, Guinsburg R, Marba ST, Martinez FE, Rugolo LM, Moreira ME, Fiori RM, Ferrari LL, Menezes JA, Venzon PS, Abdallah VQ, Duarte JL, Nunes MV, Anchieta LM, Alves Filho N. Effects of therapeutic approach on the neonatal evolution of very low birth weight infants with patent ductus arteriosus. J Pediatr (Rio J). 2014 Nov-Dec;90(6):616-23. doi: 10.1016/j.jped.2014.04.010. Epub 2014 Jul 19. PMID 25046256
- [Result] Lopez Sousa M, Perez Feal A, Soto A, Fraga JM, Couce ML. [Left vocal cord paralysis after patent ductus arteriosus surgery]. An Pediatr (Barc). 2015 Jan;82(1):e7-e11. doi: 10.1016/j.anpedi.2014.04.001. Epub 2014 May 10. Spanish. PMID 24815768
- [Result] Gimeno Navarro A, Cano Sanchez A, Fernandez Gilino C, Carrasco Moreno JI, Izquierdo Macian I, Gutierrez Laso A, Morcillo Sopena F. [Ibuprofen versus indomethacin in the treatment of patent ductus arteriosus in preterm infants]. An Pediatr (Barc). 2005 Sep;63(3):212-8. doi: 10.1157/13078483. Spanish. PMID 16219273
- [Result] Clyman RI, Chorne N. Patent ductus arteriosus: evidence for and against treatment. J Pediatr. 2007 Mar;150(3):216-9. doi: 10.1016/j.jpeds.2006.12.048. No abstract available. PMID 17307530
- [Result] Van Overmeire B, Chemtob S. The pharmacologic closure of the patent ductus arteriosus. Semin Fetal Neonatal Med. 2005 Apr;10(2):177-84. doi: 10.1016/j.siny.2004.10.003. Epub 2004 Dec 15. PMID 15701582
- [Result] Mosalli R, Alfaleh K. Prophylactic surgical ligation of patent ductus arteriosus for prevention of mortality and morbidity in extremely low birth weight infants. Cochrane Database Syst Rev. 2008 Jan 23;2008(1):CD006181. doi: 10.1002/14651858.CD006181.pub2. PMID 18254095